CLINICAL TRIAL: NCT02832778
Title: Steady-state Pharmacokinetics of Efavirenz (Sustiva/Stocrin) 400 mg Once Daily in the Presence of Rifampicin and Isoniazid (Rifinah or the Local Generics)
Brief Title: Pharmacokinetics of Efavirenz in the Presence of Rifampicin and Isoniazid
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Mylan Inc. (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT062
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: HIV
MeSH Terms: interventions — efavirenz; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine; Lamivudine; lamivudine, zidovudine drug combination; Rifampin; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage 1 London (Experimental): Stage 1, London:
  * Phase 1 (2 weeks): tenofovir/emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine plus efavirenz (Sustiva/Stocrin) 400 mg once daily
  * Phase 2 (12 weeks): tenofovir/emtricitabine or tenofovir /lamivudine or zidovudine/lamivudine) plus efavirenz (Sustiva/Stocrin) 400 mg once daily plus Rifinah or local generics once daily (rifampicin 600 mg and isoniazid 300 mg if ≥50kg or rifampicin 450 mg and isoniazid 300 mg if <50kg.)
  Interventions: Drug: Efavirenz; Drug: tenofovir /emtricitabine; Drug: tenofovir/lamivudine; Drug: lamivudine/zidovudine; Drug: Rifinah or local generics
- Stage 2 Kampala (Experimental): Tenofovir/emtricitabine or lamivudine or zidovudine/lamivudine plus efavirenz (Sustiva/Stocrin) 400 mg once daily plus Rifinah or local generics once daily (rifampicin 600 mg and isoniazid 300 mg if ≥ 50 kg or rifampicin 450 mg and isoniazid 300 mg if <50kg).
  Interventions: Drug: Efavirenz; Drug: tenofovir /emtricitabine; Drug: tenofovir/lamivudine; Drug: lamivudine/zidovudine; Drug: Rifinah or local generics

INTERVENTIONS:
Drug: Efavirenz — Efavirenz 400mg
  Other Names: Sustiva; Stocrin; Atripla
Drug: tenofovir /emtricitabine — tenofovir 245 mg/emtricitabine 200mg
Drug: tenofovir/lamivudine — tenofovir 245mg/lamivudine 300mg
Drug: lamivudine/zidovudine — lamivudine 300mg/zidovudine 600mg
Drug: Rifinah or local generics — Rifampicin 600 mg and isoniazid 300 mg if ≥50kg or rifampicin 450 mg and isoniazid 300 mg if <50kg.)
  Other Names: Rifampicin and isoniazid

SUMMARY:
The purpose of the study is to measure the drug levels in the blood of HIV-infected individuals taking anti- HIV medication efavirenz 400 mg once daily in the presence of anti-TB medication rifampicin and isoniazid. The study is being run in two-stages - London (Stage 1) and Kampala (Stage 2).

In London (Stage 1): HIV-1 infected patients (without tuberculosis infection) on established treatment with a combination based on 600 mg efavirenz dose will be recruited.

In Kampala (Stage 2): Patients with both HIV-1 and tuberculosis infection being treated with 600 mg efavirenz combination for HIV AND undergoing TB treatment with a dual therapy regimen contaning rifampicin and isoniazid will be recruited.

Efavirenz-containing regimens are recommended as first-line therapy for HIV-TB co-infected patients. It has been shown there is a lack of a significant difference between efavirenz 400 mg and efavirenz 600 mg, indicating that 400 mg efavirenz is non-inferior to the standard dose.

The advantages of antiretroviral dose reductions may translate into greater benefits for more individuals infected by HIV globally, since they may allow access programs to reach higher numbers of infected patients and compensate for the finite global manufacturing capacity and increasing demand. For efavirenz, significant price reductions have been achieved through elimination of trade, logistics and manufacturing capacity barriers, and further price reductions could be achieved with a significant reduction in the cost of pharmaceutical ingredients. However, no data on the PK and effectiveness of efavirenz 400 mg once daily during TB treatment has been produced. Given that many patients on Efavirenz- based ART will need to be treated for TB during their lifetime and rifampicin is one of the most commonly used treatment for tuberculosis, it is important to study the reduced dose under carefully monitored conditions prior to roll out of a lower dose standard treatment. Therefore, we aim to investigate the PK of efavirenz 400 mg once daily in HIV-infected individuals in the presence of rifampicin and isoniazid in London, UK and in HIV/TB-co-infected individuals on dual anti-TB treatment in Kampala, Uganda

DETAILED DESCRIPTION:
Protocol Number: SSAT 062

EudraCT Number: 2014-002608-26

Name of Investigational Product: Sustiva/Stocrin/Atripla; Rifinah or local generic 300/150 Name of active ingredients: Efavirenz/ rifampicin/ isoniazid

Study title:Steady-state pharmacokinetics of efavirenz (Sustiva/Stocrin) 400 mg once daily in the presence of rifampicin and isoniazid (Rifinah or the local generics)

Name of Non Investigational Medicinal Product: 2 nucleoside reverse transcriptase inhibitors (Tenofovir/ emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine)

Phase of study: Phase I

Objectives: The objectives of this study are:

Primary:

1. To evaluate the steady-state pharmacokinetics of efavirenz (Sustiva/Stocrin) 400 mg once daily during co-administration with rifampicin and isoniazid (Rifinah or local generic)

Secondary:

1. To assess the safety and tolerability of efavirenz (Sustiva/Stocrin) 400 mg once daily during co-administration with rifampicin and isoniazid (Rifinah or local generic)
2. To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure
3. Exploratory: To investigate the impact of anti-retroviral drugs on platelet function in people living with HIV

Study design:

Two-centre, two-stage, 98/99 days in London (Stage 1) and 28 days in Kampala (Stage 2) (excluding screening and follow up), open-label, pharmacokinetic study

Indication:

London: HIV-1 infected patients (without tuberculosis infection) on established treatment with a combination based on 600 mg efavirenz dose Kampala: Patient with both HIV-1 and tuberculosis infection being treated with 600 mg efavirenz combination for HIV AND undergoing TB treatment with a dual therapy regimen contaning rifampicin and isoniazid

Methodology:

Measurements of efavirenz concentrations and efavirenz pharmacokinetic profiles in the absence (Stage 1 only) and in the presence of rifampicin and isoniazid in two populations of HIV-infected individuals:

1. without TB (Stage 1, London)
2. with TB (Stage 2, Kampala)

Planned sample size:

Stage 1, London: For this sequential design, a sample size of 25 patients would provide at least 80% power to detect a decrease in efavirenz Cmin of 20% during the combined rifampicin/isoniazid-efavirenz phase, compared to the efavirenz alone phase.

Up to 40 subjects may be screened and enrolled to have 25 HIV-infected patients completing the study.

Stage 2, Kampala: A pilot study in 10 patients in Uganda with HIV and TB co-infection and on anti-HIV treatment and anti-TB treatment will also be performed to validate findings of the London PK study in a TB-infected population.

Up to 25 subjects may be screened and enrolled to have 10 HIV/TB-co-infected patients completing the pilot sub-study

Summary of eligibility criteria:

Stage 1, London: HIV-1 infected males or females of at least 18 years, treated with a stable efavirenz based combination regimen (tenofovir/ emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine) for at least the preceding 12 weeks and with an undetectable viral load and a CD4+ T-cell count > 100 cell/mm3.

Stage 2, Kampala: HIV-1 infected males or females of at least 18 years, treated with a stable efavirenz based combination regimen (tenofovir /emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine) for at least the preceding 12 weeks, with a CD4+ T-cell count > 100 cell/mm3, co-infected with TB and undergoing anti-TB treatment with rifampicin and isoniazid-containing regimens.

Duration of treatment:

London: 98 / 99 (+/- 1) days (excluding screening and follow up visits) Kampala: 28 days (+/- 7) days (excluding screening and follow up visits)

Dose and route of administration:

All study drugs will be administered orally to subjects with the following schedule:

Stage 1, London:

* Phase 1 (2 weeks): tenofovir/emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine plus efavirenz (Sustiva/Stocrin) 400 mg once daily
* Phase 2 (12 weeks): tenofovir/emtricitabine or tenofovir /lamivudine or zidovudine/lamivudine) plus efavirenz (Sustiva/Stocrin) 400 mg once daily plus Rifinah or local generics once daily (rifampicin 600 mg and isoniazid 300 mg if ≥50kg or rifampicin 450 mg and isoniazid 300 mg if <50kg.)

Stage 2, Kampala:

Tenofovir/emtricitabine or lamivudine or zidovudine/lamivudine plus efavirenz (Sustiva/Stocrin) 400 mg once daily plus Rifinah or local generics once daily (rifampicin 600 mg and isoniazid 300 mg if ≥ 50 kg or rifampicin 450 mg and isoniazid 300 mg if < 50kg).

Criteria for evaluation:

Stage 1, London: Pharmacokinetic (PK) parameters of efavirenz will be evaluated on blood drawn on days:

* 14/15 (2 weeks after reducing efavirenz dose from 600 mg to 400 mg)
* 42/43 (4 weeks after Rifinah or local generics initiation at start of phase 2) and
* 98/99 (12 weeks after Rifinah or local generics initiation)
* PK profile at 0 (pre-dose), 2, 4, 8, 12 and 24 hours post administered dose.

Stage 2, Kampala: Pharmacokinetic parameters of efavirenz will be evaluated on blood drawn on:

* days 28 +/- 7 days (while on anti-TB medications)
* PK profile at 0 (pre-dose), 2, 4, 8, 12 and 24 hours post last dose.

Safety and tolerability of medications will also be assessed by questioning to collect adverse event symptoms, physical examination and laboratory parameters, performed at regular intervals during the study, including efavirenz therapeutic drug monitoring (TDM) once/twice a week.

Endpoints:

Primary endpoint:

1. Steady state plasma concentrations of efavirenz when administered at 400 mg once daily in the presence of rifampicin and isoniazid

Secondary endpoints:

1. Safety and tolerability of efavirenz when administered at 400 mg once daily in the presence of rifampicin and isoniazid.
2. Relationship between genetic polymorphisms and exposure to efavirenz.
3. Exploratory: impact of anti-retroviral drugs or platelet function in people living with HIV.

ELIGIBILITY:
Inclusion Criteria - LONDON

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
2. Male or non-pregnant, non-lactating females.
3. HIV-1-infected on an antiretroviral regimen containing tenofovir, emtricitabine, lamivudine or zidovudine/lamivudine and efavirenz 600 mg once daily for at least 12 weeks.
4. With an undetectable viral load for at least 12 weeks (re-testing is allowed).
5. CD4 count >100 cells/mm3.
6. Between 18 to 60 years, inclusive.
7. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
8. Women of childbearing potential (WOCBP) must be using an adequate and effective double barrier method of contraception (appendix 4) and is willing to continue practising these birth control methods during the trial to avoid pregnancy and for a period of at least 12 weeks after the last dose of study medication. Note: Non-childbearing potential is defined as either post-menopausal (12 months of spontaneous amenorrhoea and ≥45 years) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy.

   Adequate contraception methods are:
   * Condom and spermicides
   * Condom and Intra-uterine device (IUD/IUS)
9. Heterosexually active males, must be using effective birth control methods and is are willing to continue practising these birth control methods during the trial and until the follow-up visit
10. TB negative according to the results of the ELISPOT testing (in case of history of treated TB, ELISPOT results can be positive).

Inclusion Criteria - KAMPALA

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
2. Male or non-pregnant, non-lactating females.
3. HIV-1-infected on an antiretroviral regimen containing 2 NRTIs plus efavirenz 600 mg once daily for at least 3 weeks.
4. With a TB diagnosis and currently undergoing anti-TB treatment with rifampicin and isoniazid-containing regimens.
5. CD4 count >100 cells/mm3.
6. Between 18 to 60 years, inclusive.
7. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
8. Women of childbearing potential (WOCBP) must be using an adequate double method of contraception to avoid pregnancy throughout the study and for a period of at least 12 weeks after the last dose of study medication

   Adequate contraception methods are:
   * Condom and spermicides
   * Condom and Intra-uterine device (IUD/IUS)
9. Heterosexually active males, must be using effective birth control methods and are willing to continue practising these birth control methods during the trial and until the follow-up visit

Exclusion criteria - LONDON

1. Any significant acute or chronic medical illness that in the opinion of the investigator may influence the study results or patient safety.
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations that in the opinion of the investigator may compromise participation into the study
3. Hepatic transaminases (AST and ALT) > Grade 1 [1.25-2.5 x upper limit of normal (ULN)].
4. Positive blood screen for hepatitis B surface antigen and/or positive hepatitis C PCR.
5. Clinically relevant alcohol or drug use (positive urine drug screen - cannabis is allowed) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events.
6. Exposure to any investigational drug or placebo within one month of first dose of study drug
7. Use of any other drugs (unless approved by the Investigator - see section 5.2), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Investigator as known not to interact with study drugs.
8. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period (See inclusion criteria number 8).
9. Heterosexual males without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period. (See inclusion criteria number 9).

Exclusion criteria - KAMPALA

1. Any significant acute or chronic medical illness (with the exception of TB) that in the opinion of the Investigator may affect the study results or patient safety (including other AIDS events)
2. Evidence of severe organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations that on the opinion of the investigator may compromise participation into the study.
3. Positive blood screen for hepatitis B surface antigen or hepatitis C antibodies.
4. History of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events.
5. Exposure to any investigational drug or placebo within one month of first dose of study drug.
6. Use of any other drugs (unless approved by the Investigator - see section 5.2), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
7. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period (see inclusion criteria number 8).
8. Heterosexual males without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period (See inclusion criteria number 9 and appendix 4).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-11-21 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Steady- state plasma concentrations of efavirenz (Sustiva/Stocrin) when administered at 400 mg once daily in the presence of rifampicin and isoniazid (Rifinah or local generics). | 127 days
  The primary endpoint will be the comparison of efavirenz (Sustiva/Stocrin) Ctrough during combined treatment with efavirenz and rifampicin/isoniazid treatment for tuberculosis, versus efavirenz (Sustiva/Stocrin) treatment alone. The efavirenz (Sustiva/Stocrin) Ctrough from each patient will be compared between the two phases using geometric mean ratios (log10 transformed data). For this sequential design, a sample size of 25 patients would provide at least 80% power to detect a decrease in efavirenz Ctrough of 20% during the combined rifampicin/isoniazid-efavirenz (Sustiva/Stocrin) phase, compared to the efavirenz alone phase. This calculation assumes two-sided testing with a 5% significance level and a within-patient coefficient of variation in efavirenz levels of no more than 30%.

SECONDARY OUTCOMES:
Safety and tolerability of efavirenz when administered at 400 mg once daily in the presence of rifampicin and ison | 127 days
  Safety and tolerability of medications will also be assessed by questions, physical examination, laboratory parameters and the DAIDS table for grading the severity of adult and pediatric adverse events. These will be performed at regular intervals during the drug study.
Relationship between genetic polymorphisms and exposure to efavirenz in order to understand whether polymorphism of certain genes encoding for efavirenz metabolic enzymes are behind differences in efavirenz pharmacokinetics between people | 127 days
  A candidate gene approach will be utilised to examine loci of interest. This procedure will provide potentially important information on genetic influences on plasma drug concentrations and give insight into how to improve the management of HIV-infected patients by individualising therapy. These studies will not be powered for genetic associations but will
  - Page 5 of 6 - enable us to build a data base of genotype-phenotype. Prospective genetic studies would need to be planned based on these preliminary data.
Exploratory: impact of anti-retroviral drugs or platelet function in people living with HIV. | 127 days
  To look at platelet function during antiretroviral intake in HIV positive individuals who take part in clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MBBS,MD,PhD, Principal Investigator — St. Stephen's AIDS Trust; Mohammed Lamorde, MBBS,MRCP,PhD, Principal Investigator — Infectious Diseases Institute
Locations (2):
- Infectious Diseases Insitute, Kampala, P.O. Box 22418, Uganda
- Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cerrone M, Wang X, Neary M, Weaver C, Fedele S, Day-Weber I, Owen A, Hill A, McClure M, Boffito M. Pharmacokinetics of Efavirenz 400 mg Once Daily Coadministered With Isoniazid and Rifampicin in Human Immunodeficiency Virus-Infected Individuals. Clin Infect Dis. 2019 Jan 18;68(3):446-452. doi: 10.1093/cid/ciy491. PMID 30084943
- See also: UNAIDS is the leading advocate for worldwide action against HIV/AIDS. It promotes partnerships among and between other UN agencies, governments, corporations, media, sports and religious organizations, community-based groups — http://www.unaids.org
- See also: BHIVA (the British HIV Association) is an organisation that represents healthcare professionals working in HIV in the UK. Its guidelines set out the medical and other care people living with HIV can expect to receive in the UK — http://www.bhiva.org